CLINICAL TRIAL: NCT01348646
Title: Adult Follow-up of Preventive Study With Brief Smoking Intervention for Adolescents
Acronym: TuNAMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: Medical Research Fund of the Tampere University Hospital, Finland (Other)
Responsible Party: Aila Kätkä, Tiedetoimikunta/PSHP:n tiedekeskus
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R08017
Record Dates: First submitted 2011-05-04; First posted 2011-05-05 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-05

CONDITIONS: Smoking
Keywords: Smoking; Adolescence; Brief intervention
MeSH Terms: conditions — Smoking | interventions — Crisis Intervention

ARMS (1):
- Lifestyle counseling (Other)
  Interventions: Behavioral: Brief intervention

INTERVENTIONS:
Behavioral: Brief intervention — The adolescents were shown a series of photographs of discoloured teeth caused by smoking. Then a mirror was given to the adolescent to let him/her see if similar stains could be seen on his/her teeth. Non-smoking adolescents also received positive feedback for being non-smokers. Duration of a single brief intervention was 2-3 minutes.

SUMMARY:
The purpose of this study was to see whether a brief intervention given in adolescence has an effect on smoking in adulthood. The investigators also wanted to clarify the significance of some known psychosocial risk factors of smoking in adulthood.

ELIGIBILITY:
Inclusion Criteria:

* Born on 1979.
* Living in Vaasa, Pietarsaari, Kokkola or Seinäjoki at school age.

Exclusion Criteria:

* Other year of birth.

Ages: 12 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2582 (Actual)
Dates: Start 2008-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
being a smoker | 29 years

SECONDARY OUTCOMES:
state of dental health | 29 years
  Decayed Missing and Filled Teeth (DMFT, DMF), Decayed teeth (DT, D), Community Periodontal Index of Treatment Need (CPITN, CPIN)
daily smoking | 15 years
amount of cigarettes smoked | 29 years
smoking mother | 15 years
smoking father | 15 years
smoking sister | 15 years
smoking brother | 15 years
smoking best friend | 15 years
smoking best friend | 29 years
willingness to experiment with smoking | 15 years
self-perceived health | 29 years
asthma diagnosis | 29 years
recurrent airway tract infections | 29 years
self esteem | 15 years
  A 10-step questionnaire
smoking time | 29 years
received 1-4 brief interventions at school age (Yes/No) | 12-15 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General Practice, Medical School, University of Tampere, Finland, Tampere, Pirkanmaa, Finland

REFERENCES:
- [Derived] Saari AJ, Kentala J, Mattila KJ. The smoking habit of a close friend or family member--how deep is the impact? A cross-sectional study. BMJ Open. 2014 Feb 18;4(2):e003218. doi: 10.1136/bmjopen-2013-003218. PMID 24549158
- [Derived] Saari AJ, Kentala J, Mattila KJ. Long-term effectiveness of adolescent brief tobacco intervention: a follow-up study. BMC Res Notes. 2012 Feb 16;5:101. doi: 10.1186/1756-0500-5-101. PMID 22339943